CLINICAL TRIAL: NCT04407858
Title: Insuffisance Cardiaque Sous Carfilzomib: étude Prospective
Brief Title: Cardiovascular Complications of Carfilzomib
Acronym: ICARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Mariana Mirabel, Associate Professor, European Georges Pompidou Hospital
Other Study IDs: 00011928 ICARE
Record Dates: First submitted 2020-05-14; First posted 2020-05-29 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Myeloma; Heart Failure; Hypertension
Keywords: Adverse drug event
MeSH Terms: conditions — Neoplasms, Plasma Cell; Heart Failure; Hypertension; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular toxicity of carfilzomib, a last generation proteasome inhibitor, is highly incident according to retrospective data. Prospective cohort study of patients initiated on carfilzomib.

ELIGIBILITY:
Inclusion Criteria:

* Intention to treat by Carfilzomib

Exclusion Criteria:

* History of carfilzomib treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort of patients starting carfilzomib treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-05-21 (Estimated); Study Completion 2022-05-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardio-vasculo-toxicity of carfilzomib | 6 months
  Number of patients with cardio-toxicity (composite endpoint) in a cohort of patients referred to a cardio-oncology before initiation of carfilzomib.

SECONDARY OUTCOMES:
Systemic hypertension | 6 months
  Number of patients with as systemic hypertension
Heart Failure Reduced Ejection Fraction | 6 months
  Number of patients with Heart Failure and Reduced Ejection Fraction
Heart Failure Preserved Ejection Fraction | 6 months
  Number of patients with Heart Failure and Preserved Ejection Fraction
Predictors of Cardiotoxicity | 6 months
  Correlation between cardio-vascular toxicity and patients' chacateristics.
Impact on outcomes | 1 year
  Compare outcomes (mortality) in patients with cardiotoxicity and no cardiotoxicty.
Safety | 1 year
  Compare outcomes (mortality) in patients with cardiotoxicity according to the continuation of carflzomib or its withdrawl.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Mirabel, Principal Investigator — Assistance Publique Hôpitaux de Paris - Université de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - Centre Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided